CLINICAL TRIAL: NCT01936896
Title: Alpha-1 Anti-Trypsin (AAT) to Quench the Acute Inflammatory Response in ST-segment Elevation Acute Myocardial Infarction
Brief Title: Alpha-1 Anti-Trypsin (AAT) Treatment in Acute Myocardial Infarction
Acronym: VCU-Alpha1RT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM15342
Record Dates: First submitted 2013-08-30; First posted 2013-09-06 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-01

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction; Heart Failure; Inflammation
MeSH Terms: conditions — Heart Failure; Inflammation | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alpha-1 anti-trypsin (AAT) (Experimental): We will use plasma derived AAT 60 mg/Kg, single infusion, within 12 hours of hospital admission for ST-segment elevation myocardial infarction (STEMI)
  Interventions: Drug: Alpha 1-Antitrypsin

INTERVENTIONS:
Drug: Alpha 1-Antitrypsin
  Other Names: Prolastin C; Aralast NP

SUMMARY:
Acute myocardial infarction is characterized by an intense inflammatory response.

The degree of the response influences clinical outcome, with 'more' inflammation promoting heart failure. In this study we plan to determine whether treatment with plasma derived alpha-1 antitrypsin will quench the inflammatory response in patients with acute ST-segment elevation myocardial infarction (STEMI).

ELIGIBILITY:
Inclusion Criteria:

* Acute STEMI defined as chest pain (or equivalent) with an onset within 12 hours and ECG evidence of ST segment elevation (>1 mm) in 2 or more anatomically contiguous leads that is new or presumably new
* Planned or completed coronary angiogram for potential intervention
* Age>21

Exclusion Criteria:

* Inability to give informed consent
* Hemodynamic instability as defined as need for inotropic or vasoactive agents, or need for mechanical support devices (including intra-aortic balloon pump)
* Pregnancy
* Preexisting congestive heart failure (American Heart Association/American College of Cardiology class C-D, New York Heart Association III-IV)
* Preexisting severe left ventricular dysfunction (EF<20%)
* Preexisting severe valvular heart disease
* Known active infections (acute or chronic)
* Recent (<14 days) or active use of anti-inflammatory drugs (not including NSAIDs or corticosteroids used for IV dye allergy only)
* Known chronic inflammatory disease (including but not limited to rheumatoid arthritis, systemic lupus erythematosus)
* Known active malignancy of any type, or prior diagnosis in the past 10 years
* Anticipated need for cardiac or major surgery
* Known active cancer (or prior diagnosis of cancer within the past 10 years)
* Known Immunoglobulin A (IgA) deficiency

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Abbate, MD, PhD, Principal Investigator — Virginia Commonwealth University; Benjamin Van Tassell, PharmD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Abouzaki NA, Christopher S, Trankle C, Van Tassell BW, Carbone S, Mauro AG, Buckley L, Toldo S, Abbate A. Inhibiting the Inflammatory Injury After Myocardial Ischemia Reperfusion With Plasma-Derived Alpha-1 Antitrypsin: A Post Hoc Analysis of the VCU-alpha1RT Study. J Cardiovasc Pharmacol. 2018 Jun;71(6):375-379. doi: 10.1097/FJC.0000000000000583. PMID 29634656

RESULTS

PARTICIPANT FLOW:
Groups:
- Alpha-1 Anti-trypsin (AAT): Plasma derived Alpha 1-Antitrypsin (AAT) 60 mg/Kg, single infusion, within 12 hours of hospital admission for ST-segment elevation myocardial infarction (STEMI)
Period: Overall Study
Arm/Group | Alpha-1 Anti-trypsin (AAT)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Alpha-1 Anti-trypsin (AAT): Plasma derived (Alpha 1-Antitrypsin) AAT 60 mg/Kg, single infusion, within 12 hours of hospital admission for ST-segment elevation myocardial infarction (STEMI)
Arm/Group | Alpha-1 Anti-trypsin (AAT)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 52.5 [33 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: C Reactive Protein (Area Under the Curve)
Description: A single area under the curve (AUC) calculation based upon C-reactive protein (CRP) values drawn at baseline, 3 days, and 14 days.
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: mg/L
Groups:
- Alpha-1 Anti-trypsin (AAT): Plasma derived AAT 60 mg/Kg, single infusion
Arm/Group | Alpha-1 Anti-trypsin (AAT)
Number analyzed (Participants) | 10
mg/L | 75.9 [31.4 to 147.8]

2. Secondary Outcome: Left Ventricular End-systolic Volume Change
Description: We will calculate the interval change between admission and 3 months in left ventricular end-systolic volume, using echocardiography
Time Frame: 3 months
Population: Only 5 patients had paired (i.e. baseline and 3 months) echocardiograms for evaluation
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Alpha-1 Anti-trypsin (AAT)
Number analyzed (Participants) | 5
mL | 2 [-6 to 19]

3. Other Pre Specified Outcome: Safety
Description: We will record the number of participants with all adverse events (cardiac and non-cardiac) over the 3 months, including infusion reactions and drug-related issues.
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Alpha-1 Anti-trypsin (AAT)
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha-1 Anti-trypsin (AAT) (N=10)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sudden death (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No